CLINICAL TRIAL: NCT05162443
Title: Expanded Access Use of Adagrasib (MRTX849) for the Treatment of Patients With Advanced Solid Tumors With a KRAS G12C Mutation
Brief Title: Expanded Access of Adagrasib (MRTX849) in Patients With Advanced Solid Tumors Who Have a KRAS G12C Mutation
Status: Approved for marketing | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA239-0067; 849-EAP-001 (Other: Mirati Protocol ID)
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; Metastatic Cancer; Malignant Neoplasm
Keywords: adagrasib; expanded access
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — adagrasib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: adagrasib (MRTX849) — adagrasib (MRTX849) will be administered orally twice daily in a continuous regimen

SUMMARY:
The objective of this EAP is to provide expanded access of adagrasib (MRTX849) to patients with previously treated advanced solid tumors harboring a KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of an advanced/metastatic solid tumor
* Confirmed presence of a KRASG12C mutation
* Ineligible for an ongoing clinical trial of MRTX849
* No available or not eligible for standard of care treatment
* Adequate organ function
* CNS Metastases (within set parameters) are allowed
* ECOG performance status of ≤ 2

Exclusion Criteria:

* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions likely to alter absorption of MRTX849 treatment or result in inability to swallow
* Prior therapy targeting a KRAS G12C mutation
* Other active cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (11):
  - California Pacific Medical Center, San Francisco, California
  - Providence Medical Group Santa Rosa - Cancer Center, Santa Rosa, California
  - Hartford Hospital, Hartford, Connecticut
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Renown Health, Reno, Nevada
  - Lehigh Valley Cancer Institute, Allentown, Pennsylvania
  - Lumi Research, Kingwood, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Seattle Integrative Cancer Center, Renton, Washington
  - Swedish Cancer Institute, Seattle, Washington

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx